CLINICAL TRIAL: NCT00931541
Title: A Phase I, Single Centre, Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability and Pharmacokinetics of Oral AZD6088 After Single Ascending Doses in Healthy Male and Non-Fertile Female Volunteers
Brief Title: AZD6088 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: D0840C00007; EudraCT N0. 2008-007936-17
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Volunteers
Keywords: Safety; Tolerability; Healthy
MeSH Terms: interventions — AZD6088

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): AZD6088 oral solution
  Interventions: Drug: AZD6088
- B (Experimental): Placebo oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6088 — Oral solution. Each subject will receive a single-dose of AZD6088.
  Arms: A
Drug: Placebo — Oral solution. Each subject will receive a single-dose of placebo.
  Arms: B

SUMMARY:
The aims of the study are to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of AZD6088 following single ascending dose administration in healthy male and non-fertile females.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male and non-fertile female healthy volunteers aged ≥18 to ≤55 years with suitable veins for cannulation or repeated venipuncture.
* Clinically normal physical findings including supine BP, pulse rate, ECG and laboratory assessments in relation to age, as judged by the investigator.
* Normal and suitable EEG, as judged by a neurologist

Exclusion Criteria:

* History of any clinically significant disease or disorder which for instance includes CNS disorder or CV disorder.
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator.
* Any clinically important abnormalities in the ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety variables (vital signs, ECG, EEG, safety laboratory values, body temp) | Sampling occasions during all visits.

SECONDARY OUTCOMES:
Pharmacokinetics | Intense PK-sampling during 3 pre-defined study days for PK profiling.
Pharmacodynamics | Sampling occasions during 3 pre-defined study days.

CONTACTS AND LOCATIONS:
Overall Officials: Biljana Lilja, Study Director — AstraZeneca R&D, Södertälje, Sweden; Marianne Kasti, Principal Investigator — Quintiles GDRU, London, UK
Locations (1):
- Research Site, London Bridge, Greater London, United Kingdom